CLINICAL TRIAL: NCT05333549
Title: Istradefylline for Parkinson Disease Cognitive Impairment
Brief Title: Istradefylline for Parkinson Disease With Cognitive Impairment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Kyowa Kirin, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HM20022119
Record Dates: First submitted 2022-04-11; First posted 2022-04-19 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Parkinson Disease; Cognitive Impairment
MeSH Terms: conditions — Parkinson Disease; Cognitive Dysfunction

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Usual care plus istradefylline (Experimental): Participants will receive usual care, and in addition, will be asked to take istradefylline daily for 26 weeks.
  Interventions: Drug: Istradefylline medication

INTERVENTIONS:
Drug: Istradefylline medication — 2 weeks on istradefylline 20mg daily, 2 weeks on istradefylline 40mg with the ability to adjust other antiparkinsonian medications, and 22 weeks on istradefylline 40mg and stable antiparkinsonian medications

SUMMARY:
The purpose of this research study is to determine whether istradefylline improves cognition in individuals with Parkinson disease with cognitive impairment.

DETAILED DESCRIPTION:
Istradefylline has been approved by the U. S. Food and Drug Administration (FDA) to reduce "off" episodes in Parkinson disease. The period when levodopa has a positive effect on Parkinson's symptoms is called on-time. Once the medication stops working, a so called "off" episode starts, where symptoms recur. Usual care for treatment of Parkinson disease with cognitive impairment is use of cognition enhancing medications also called cholinesterase inhibitors. In this study, participants will receive usual care, and in addition, they will be asked to take istradefylline daily for 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Meet criteria for probable Parkinson disease dementia or PD-MCI (mild cognitive impairment)
* Age greater than 50
* Hoehn and Yahr stage < 4 in "on" state
* Currently taking carbidopa/levodopa
* Antiparkinsonian medications stable for at least 4 weeks prior to baseline visit
* Cholinesterase inhibitor dose stable for 8 weeks prior to baseline visit

Exclusion Criteria:

* Meet criteria for dementia with Lewy bodies, including dementia onset prior to or within 1 year of parkinsonism onset
* Presence of troublesome dyskinesias
* Pregnancy or possibility of becoming pregnant during the study period.
* Moderate or severe hepatic impairment
* dementia too severe to complete study measures or to adhere to medication schedule

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2025-06-09 (Actual); Study Completion 2025-06-09 (Actual)

PRIMARY OUTCOMES:
Change in executive function - Card Sort test | Baseline to 26 weeks
  Executive function will be assessed using the Card Sort Test from the NIH Toolbox Cognition Battery. Participants will be assessed at baseline, 4 weeks, 14 weeks, and 26 weeks

SECONDARY OUTCOMES:
Change in neurocognitive outcomes | Baseline to 26 weeks
  NIH Toolbox Cognition Battery (NTCB) consists of multiple self-report and clinician reported tests. The assessments can be completed on a tablet device and a composite as well as sub-scores are calculated. Higher scores are indicative of better functioning. Participants will be assessed at baseline, 4 weeks, 14 weeks, and 26 weeks.
Change in recall | Baseline to 26 weeks
  Immediate and delayed recall will be assessed using the Hopkins Verbal Learning Test - Revised, which will be administered by a trained clinician. Higher scores indicate better recall. Participants will be assessed at baseline, 4 weeks, 14 weeks, and 26 weeks.
Change in oral fluency | Baseline to 26 weeks
  In the Controlled Oral Word Association Test (FAS, animals) (COWAT) the participant is asked to make verbal associations to different letters of the alphabet by saying all the words which they can think of beginning with a given letter. Higher scores indicate better oral fluency. Participants will be assessed at baseline, 4 weeks, 14 weeks, and 26 weeks.
Change in executive function - Trail Making Test | Baseline to 26 weeks
  Participants will complete the Trail Making Test (TMT) which is a timed test of executive function. Scores are the number of seconds needed to complete the test with higher scores indicate poorer executive function. Participants will be assessed at baseline, 4 weeks, 14 weeks, and 26 weeks.
Change in cognitive status | Baseline to 26 weeks
  Participant's cognitive status will be assessed using the Montreal Cognitive Assessment score. Higher scores indicated better cognitive status. Participants will be assessed at baseline, 4 weeks, 14 weeks, and 26 weeks.
Change in higher cortical functions | Baseline to 26 weeks
  The Dementia Rating Scale-2 (DRS-2) measures deficits in a large range of higher cortical functions and differentiates deficits of varying severity levels. The DRS-2 yields five subscales as well as an overall cognitive functioning score. Higher scores higher impairment. Participants will be assessed at baseline, 4 weeks, 14 weeks, and 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Barrett, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No